CLINICAL TRIAL: NCT06773455
Title: A Single-Center, Open-Label Study to Evaluate Tralokinumab in Atopic Dermatitis Subjects Who Experienced Inadequate Response on Dupilumab
Brief Title: Tralokinumab for Dupilumab Failures
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Psoriasis Treatment Center of Central New Jersey (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETC05
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — tralokinumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tralokinumab (Experimental)
  Interventions: Drug: tralokinumab

INTERVENTIONS:
Drug: tralokinumab — 600mg at week 0 followed by 300mg Q2W for 24 weeks

SUMMARY:
24-week study of 20 atopic dermatitis patients who have been treated with dupilumab will receive Tralokinumab 600mg at week 0 followed by 300mg Q2W for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult ≥ 18 years of age;
* All participants must have prior treatment with dupilumab for atopic dermatitis meeting one of the following conditions:

  * Participants who stopped dupilumab treatment due to non-response, partial response, loss of efficacy must have been previously treated with dupilumab for at least 12 weeks.
  * Participants who stopped dupilumab treatment due to intolerance or AEs to the drug may enter the study with no required prior length of dupilumab treatment. AE's must be resolved prior to 1st tralokinumab dose.
* Females of childbearing potential (FCBP) must have a negative urine pregnancy test at Baseline. FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options: hormonal contraception; intrauterine device (IUD); tubal ligation; or partner's vasectomy; Male or female condom diaphragm with spermicide, cervical cap with spermicide, or contraceptive sponge with spermicide.

Subject is a candidate for systemic therapy.

* Subject must be in general good health as judged by the Investigator, based on medical history, physical examination.
* Able and willing to give written informed consent prior to performance of any study-related procedures.

Exclusion Criteria:

* Subjects with previous exposure to tralokinumab.
* Known or suspected hypersensitivity to tralokinumab or any of its excipients.
* Women of childbearing potential who are pregnant, intend to become pregnant, or are lactating.
* Use of tanning beds or phototherapy within 4 weeks of baseline
* Use of systemic therapies (systemic steroids, cyclosporine, oral JAK inhibitors etc.) for atopic dermatitis within 4 weeks
* Patient non-compliant with Dupixent dosing based on investigator discretion.
* Any clinically significant (as determined by the investigator) cardiac, endocrinologic, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, immunologic disease, or other major disease that is uncontrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving IGA 0 or 1 at week 16 | 16 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Psoriasis Treatment Center of New Jersey, East Windsor, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wollenberg A, Blauvelt A, Guttman-Yassky E, Worm M, Lynde C, Lacour JP, Spelman L, Katoh N, Saeki H, Poulin Y, Lesiak A, Kircik L, Cho SH, Herranz P, Cork MJ, Peris K, Steffensen LA, Bang B, Kuznetsova A, Jensen TN, Osterdal ML, Simpson EL; ECZTRA 1 and ECZTRA 2 study investigators. Tralokinumab for moderate-to-severe atopic dermatitis: results from two 52-week, randomized, double-blind, multicentre, placebo-controlled phase III trials (ECZTRA 1 and ECZTRA 2). Br J Dermatol. 2021 Mar;184(3):437-449. doi: 10.1111/bjd.19574. Epub 2020 Dec 30. PMID 33000465
- [Background] Vangipuram R, Tyring SK. Dupilumab for Moderate-to-Severe Atopic Dermatitis. Skin Therapy Lett. 2017 Nov;22(6):1-4. PMID 29091379
- [Background] Bieber T. Atopic dermatitis. N Engl J Med. 2008 Apr 3;358(14):1483-94. doi: 10.1056/NEJMra074081. No abstract available. PMID 18385500
- [Background] Akdis CA, Akdis M, Bieber T, Bindslev-Jensen C, Boguniewicz M, Eigenmann P, Hamid Q, Kapp A, Leung DY, Lipozencic J, Luger TA, Muraro A, Novak N, Platts-Mills TA, Rosenwasser L, Scheynius A, Simons FE, Spergel J, Turjanmaa K, Wahn U, Weidinger S, Werfel T, Zuberbier T; European Academy of Allergology and Clinical Immunology/American Academy of Allergy, Asthma and Immunology. Diagnosis and treatment of atopic dermatitis in children and adults: European Academy of Allergology and Clinical Immunology/American Academy of Allergy, Asthma and Immunology/PRACTALL Consensus Report. J Allergy Clin Immunol. 2006 Jul;118(1):152-69. doi: 10.1016/j.jaci.2006.03.045. PMID 16815151
- [Background] Schmitt J, Langan S, Deckert S, Svensson A, von Kobyletzki L, Thomas K, Spuls P; Harmonising Outcome Measures for Atopic Dermatitis (HOME) Initiative. Assessment of clinical signs of atopic dermatitis: a systematic review and recommendation. J Allergy Clin Immunol. 2013 Dec;132(6):1337-47. doi: 10.1016/j.jaci.2013.07.008. Epub 2013 Sep 12. PMID 24035157

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT06773455/Prot_SAP_000.pdf